CLINICAL TRIAL: NCT00475098
Title: Effect of Low Molecular Weight Heparin on Survival of Stage I,II or IIIA Non Small Cell Lung Cancer. A Multicenter, Open, Randomized Controlled Trial.
Brief Title: Effect of Low Molecular Weight Heparin: Tinzaparin in Lung Tumours (TILT)
Acronym: TILT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051084
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: Low molecular weight heparin; Lung cancer; Non small cell lung cancer; Adjuvant therapy; Anticoagulants; Heparin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Tinzaparin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Tinzaparin sodium 100 UI/Kg/OD for 12 weeks
- B (Experimental)
  Interventions: Drug: Tinzaparin sodium 100 UI/Kg/OD for 12 weeks

INTERVENTIONS:
Drug: Tinzaparin sodium 100 UI/Kg/OD for 12 weeks — treatment in lung tumours
  Other Names: treatment in lung tumours

SUMMARY:
Experiments suggest that low molecular weight heparin (LMWH) inhibits tumor growth and metastasis. Studies in humans suggest that LMWH is associated with a higher survival in patients with cancer related thrombosis. Two recent studies suggest that LMWH may increase the survival of patients with cancer who do not have an associated thrombosis. The purpose of the study is to assess the effect of LMWH on the overall survival of patients with localized non-small cell lung cancer after complete surgical resection.

DETAILED DESCRIPTION:
Phase III, prospective, multicentric, randomized, controlled, open trial in parallel groups with a blind adjudication of all end-point criteria.

Reference therapy :

Patients randomized to the control group will receive postoperative treatment according to local practice in the participating centers. However, the participating centers will have to comply with the following guidelines.

Adjuvant chemotherapy:

Adjuvant chemotherapy will be offered in all patients with stage II and stage IIIA cancers. Adjuvant chemotherapy will be platin based and include two drugs for a maximum of 4 cycles. Each center will have to select one regimen before the beginning of the study for all patients included in the study.

Preoperative chemotherapy:

Patients who had chemotherapy before surgery can be included in the study provided that they had a complete surgical resection. In this case the tumor stage for stratification will be the pathologic stage assessed after surgery.

Stage I cancers:

Patients with stage I cancer who will not be selected for postoperative chemotherapy can be included in the study. Contraindication to chemotherapy Patients with a contraindication to postoperative chemotherapy and those who refuse chemotherapy can be included in the study provided they fulfill all inclusion and exclusion criteria.

Experimental treatment:

Experimental treatment is tinzaparin administered subcutaneously once a day at the dose of 100 IU/Kg during a twelve week period beginning after a maximum period of 8 weeks after surgery. Patients randomized in the experimental group will receive adjuvant postoperative treatment according to local practice with the same guidelines as in the control group.

* Patient follow-up:

All patients will be followed according to local practice, but at least two outpatient visits with a chest radiograph will be planned each year during the three year follow-up period after last inclusion.

* Duration of the trial:

Inclusion period (first patient in to last patient in) : 6 years. Patient total follow-up (from surgery to end of follow-up) : 3 years after last inclusion (first enrolled patients were followed 9 years). Total study period : 9 years.

ELIGIBILITY:
Inclusion Criteria:

Patients with completely resected non-small cell lung cancer of stage I, II, or IIIA T3N1 confirmed by histology can be included in the study Patients who had preoperative chemotherapy, those who are selected for adjuvant chemotherapy and those who are not candidates for adjuvant chemotherapy (because they have a contraindication to chemotherapy or they have a stage I cancer) are eligible for the study Written informed consent age > 18 years

Exclusion Criteria:

Previous heparin induced thrombocytopenia Allergy to tinzaparin Allergy to sulfites Renal failure with a creatinin clearance < 30 ml/min according to COCKROFT formula Prothrombin time < 50% Platelet count < 100 G/L Increased bleeding risk: ongoing hemorrhage, major bleeding within 10 days, previous intracerebral bleeding, uncontrolled hypertension (SAP > 180 mmHg or DAP > 120 mmHg) Indication for curative anticoagulant treatment on inclusion More than 6 weeks between surgery and inclusion Known pregnancy or no efficient contraception for women of childbearing age Breast feeding Previous malignant disease diagnosed within 2 years except in situ carcinoma of the uterine cervix or spinal-cellular or baso-cellular cutaneous carcinoma Inclusion in another therapeutic trial at the time of inclusion Treatment with an experimental drug within 30 days before inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2007-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall 3-year mortality | overall 3-years
  The first included patients will be followed 9 years with no impact on the total duration of the study.

SECONDARY OUTCOMES:
Major bleeding time | Overall five year survival
  Disease free survival of the first enrolled patients will be assessed 9 years after inclusion
Symptomatic venous thromboembolic events | Overall five year survival
  Symptomatic venous thromboembolic events of the first enrolled patients will be assessed 9 years after inclusion
Cancer related mortality | Overall five year survival
  Cancer related mortality of the first enrolled patients will be assessed 9 years after inclusion
Disease free survival | Overall five year survival
  Disease free survival of the first enrolled patients will be assessed 9 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Result] Alifano M, Benedetti G, Trisolini R. Can low-molecular-weight heparin improve the outcome of patients with operable non-small cell lung cancer? An urgent call for research. Chest. 2004 Aug;126(2):601-7. doi: 10.1378/chest.126.2.601. No abstract available. PMID 15302749
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Meyer G, Besse B, Doubre H, Charles-Nelson A, Aquilanti S, Izadifar A, Azarian R, Monnet I, Lamour C, Descourt R, Oliviero G, Taillade L, Chouaid C, Giraud F, Falcoz PE, Revel MP, Westeel V, Dixmier A, Tredaniel J, Dehette S, Decroisette C, Prevost A, Pichon E, Fabre E, Soria JC, Friard S, Stern JB, Jabot L, Dennewald G, Pavy G, Petitpretz P, Tourani JM, Alifano M, Chatellier G, Girard P. Anti-tumour effect of low molecular weight heparin in localised lung cancer: a phase III clinical trial. Eur Respir J. 2018 Oct 4;52(4):1801220. doi: 10.1183/13993003.01220-2018. Print 2018 Oct. PMID 30262574